CLINICAL TRIAL: NCT06013215
Title: PULSE - Paramètres de l'Impulsion électrique et Population Neuronale Chez le Patient implanté cochléaire - Etude en Ouvert, Non contrôlé, Non randomisée
Brief Title: Electrical Impulse Parameters and Neuronal Population in the Cochlear Implanted Patient-PULSE
Acronym: PULSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DR230050-PULSE; 2023-A00476-39 (Other: ANSM); DR230050 (Registry Identifier: Promoter ID)
Record Dates: First submitted 2023-07-27; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Sensorineural Hearing Loss
Keywords: hearing loss; cochlear implant; psychoacoustic; charge integration efficiency
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cochlear implant users with Neuro Zti array (Experimental): Post-lingually cochlear implant users with 12 months of auditory experience Modifications of pulse parameters to determine the charge integration efficiency which is related with neuron survival population
  Interventions: Other: Cochlear implant (Oticon) stimulation parameter optimization

INTERVENTIONS:
Other: Cochlear implant (Oticon) stimulation parameter optimization — The pulse amplitude and/or the pulse phase duration will be optimize to improve the intensity resolution of the cochlear implant which may benefit speech perception

SUMMARY:
The cochlear implant provides good auditory performance despite high inter-individual variability, but performance in noise remains limited. Modification of the coding strategies could improve these performances. A better characterization of the remaining neuronal population by looking for the charge integration efficiency (which depends on the duration and the amplitude of the electrical pulse) would allow an optimization of the settings by adapting either the duration or the amplitude of the pulse according to the quality of the remaining neuronal population.

DETAILED DESCRIPTION:
The cochlear implant provides good auditory performance despite high inter-individual variability, but performance in noise remains limited. Modification of the coding strategies could improve these performances. Currently, the intensity perceived by the patient is coded by the duration and the amplitude of the electrical impulse but companies have different approaches and fix one of the two parameters for the setting of the processors. A better characterization of the remaining neuronal population by looking for the charge integration efficiency (which depends on the duration and the amplitude of the electrical pulse) would allow an optimization of the settings by adapting either the duration or the amplitude of the pulse according to the quality of the remaining neuronal population.

ELIGIBILITY:
Inclusion Criteria:

* post-lingually deaf adults with at least one year of cochlear implant experience
* unilateral and bilateral cochlear implant recipients
* Oticon device with Neuro Zti array
* Patient affiliated to french social security
* Consent signed

Exclusion Criteria:

* Patients under court protection, guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Calculate the charge integration efficiency along the electrodes | 4 hours
  Charge integration efficiency will be determined for each electrode by noting the minimum and maximum loudness perceived by the patient as function of pulse phase duration and amplitude

SECONDARY OUTCOMES:
Questionnaire between Intensity discrimination and charge integration efficiency | 4 hours
  3 electrodes that span the range of charge integration efficiency values will be selected as test electrodes. Three intensities will be presented to the patient through the implant and it will be asked to the patient to determine which intensity is higher than the others.

CONTACTS AND LOCATIONS:
Overall Officials: David Bakhos, Principal Investigator — University Hospital, Tours